CLINICAL TRIAL: NCT02183857
Title: Femoral Arterial Cannulation Performed by Residents: A Comparison Between Ultrasound-Guided and Landmark Technique in Infants and Children Undergoing Cardiac Surgery
Brief Title: Ultrasound-Guided vs Landmark Technique for Femoral Arterial Cannulation in Pediatric Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Sahar Sayyid, Professor, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ANES.SS.12
Record Dates: First submitted 2014-07-03; First posted 2014-07-08 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Time Needed to Achieve a Successful Cannulation of the Femoral Artery in Pediatric Cardiac Surgery
Keywords: children; congenital heart disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound (Other): Patients in group Ultrasound will have their femoral arterial lines inserted under the guidance of US. The Ultrasound equipment used is a SonoSite 180 PLUS with an L25/10- to 5-MHz linear array transducer (SonoSite, Inc., Bothell, WA)
  Interventions: Device: Ultrasound
- Landmark (Other): No Device is used. Patients in group Landmark will have their femoral line inserted using the blinded, external landmark-guided technique. After localization of the femoral artery by identifying the pulse in the femoral triangle immediately distal to the inguinal ligament.
  Interventions: Other: Landmark

INTERVENTIONS:
Device: Ultrasound
  Other Names: SonoSite 180 PLUS
  Arms: Ultrasound
Other: Landmark
  Arms: Landmark

SUMMARY:
The use of ultrasound guidance by senior residents learning the technique of femoral artery catheterization is superior to the landmark technique.

DETAILED DESCRIPTION:
The insertion of percutaneous femoral catheter is the method of choice for arterial monitoring in pediatric patients undergoing cardiac surgery at American University of Beirut Medical Center. It is easier to access since it is a bigger vessel and matches better the aortic pressure immediately post initiation of bypass than the radial artery. Utilizing ultrasound in radial artery cannulation has been well described (1). A meta-analysis of 4 trials showed that, ultrasound guidance for radial artery catheterization improved first-pass success rate compared to the palpation method (2). Two of these trials were for pediatric patients where in one study ultrasound-guided radial arterial cannulation in 30 small children improved success rate with fewer attempts required with the ultrasound technique than with the traditional technique (3). However, in another study of 152 children under 12 years of age requiring radial artery cannulation, there were no statistically significant differences between the groups in time to successful cannulation, total number of attempts, number of successful cannulations during the first attempt, or in the number of cannulae used for catheterization (4). No previous study compared the use of ultrasound guidance vs landmark for femoral artery cannulation in the pediatric age group in particular for the teaching of anesthesia residents.

The hypothesis is that the use of ultrasound guidance by senior residents learning the technique of femoral artery catheterization is superior to the landmark technique.

The investigators will design a prospective randomized trial to compare the use of ultrasound guidance versus landmark technique in 110 children undergoing cardiac surgery. The inclusion criteria are ASA III or IV children under 12 years of age. Exclusion criteria are hematoma or infections at the potential site of insertion, need for emergency surgery, and hemodynamic instability.

The risks to subjects include no more than the usual risks of arterial cannulation (infection and hematoma formation). Adverse events will be monitored, reported and treated appropriately.

Privacy and confidentiality will be respected. Data will be kept under lock with the primary investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Infants and children under 12 years of age.
2. American Society of Anesthesiologist Physical Status (ASA) III or IV.
3. Patients with congenital heart disease undergoing cardiac surgery who do not have existing arterial line access.
4. Parents/guardians/patients willing to sign consent.

Exclusion Criteria:

1. Hematoma or infections at the potential site of insertion.
2. Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.
3. Need for emergency surgery.
4. Hemodynamic instability

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
the time needed to achieve a successful cannulation of the femoral artery. | The time to successful cannula insertion will be calculated from the time of skin penetration until proper placement of the catheter is confirmed by an arterial waveform seen on the monitor after connecting the catheter to a transducer

CONTACTS AND LOCATIONS:
Overall Officials: Sahar M Siddik-Sayyid, MD, Principal Investigator — AUBMC
Locations (1):
- American University of Beirut Medical center, Beirut, Lebanon